CLINICAL TRIAL: NCT06344585
Title: Drop-out of Infertile Couples: a Prospective Study in Which Dropout Women in 2021 Were Enrolled to Answer to a Questionnaire Exploring Their Reasons and a Retrospective Study Which Explored the Factors for Dropout Over 10 Years
Brief Title: Drop-out of Infertile Couples: a Large Single Center Experience Over 10 Years
Acronym: dropout
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: DROPOUT
Record Dates: First submitted 2024-03-27; First posted 2024-04-03 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Infertility
Keywords: infertility; dropout
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Drop out: Women who had their first access from 2012 to 2021 and never returned back
  Interventions: Other: Drop out patients who had their first access in 2021 were additionally asked to answer to a phone -call questionnaire to assess their motivation of discontinuation
- Non drop out: Women who had their first access from 2012 to 2021 and returned back for subsequent treatment

INTERVENTIONS:
Other: Drop out patients who had their first access in 2021 were additionally asked to answer to a phone -call questionnaire to assess their motivation of discontinuation — A prospective comprehensive analysis of the data contained within patient charts, encompassing personal histories and demographic details, was extracted from the internal database of the Humanitas Fertility Center. This analysis aimed at elucidating the individual reasons for treatment discontinuation after the initial clinical visit throughout the year 2021. Additionally a tailored questionnaire was administered to patients via telephone by a member of Humanitas Fertility Center staff in July 2023.
  The questionnaire was submitted to the patients via a phone call. The questionnaire comprised nine questions with response limited to 'Yes' and 'No' options for all queries.
  Groups: Drop out

SUMMARY:
Conducted at a single-center, this prospective-retrospective study focused on all couples who initiated their journey at the Fertility Center of Humanitas Research Hospital, Rozzano (Milan), Italy.

The prospective study focused on the couples whose first consultation occurred in 2021. A tailored questionnaire was administered via telephone by staff members to gather insights into the personal reasons for treatment discontinuation among non-returning patients.

Conversely, the retrospective study included all infertile couples initiating treatment between January 2012 and December 2021 at the Fertility Center. Data encompassing personal history and demographic details were extracted from the internal database of Humanitas Fertility Center to assess the factors involved in a treatment discontinuation.

DETAILED DESCRIPTION:
Background In recent years refinements and improvements in In vitro Fertilization and embryo transfer (IVF-ET) techniques have significantly enhanced the efficacy of infertility treatments, offering renewed hope to countless couples struggling with conception. Simultaneously, there has been a notable surge in the number of couples seeking IVF procedures. Studies indicate that, under optimal conditions, approximately 83% of women undergoing IVF treatment could achieve a live birth within eight complete cycles, a rate comparable to natural conception among fertile non-contraceptive users. Despite these encouraging statistics, a significant portion of couples discontinue treatment prematurely.

Objectives The study aims at evaluating the dropout rate among couples following their first access to the Fertility Center. It seeks to elucidate the concept of treatment continuation versus dropout and to identify the determinants influencing these decisions among infertile couples. Additionally, the study aims at investigating the factors contributing to non-return among patients who did not proceed with further treatment.

Materials and methods Conducted at a single-center, this prospective-retrospective study focused on all couples who initiated their journey at the Fertility Center of Humanitas Research Hospital, Rozzano (Milan), Italy.

The prospective study focused on the couples whose first consultation occurred in 2021. A tailored questionnaire was administered via telephone by staff members to gather insights into the personal reasons for treatment discontinuation among non-returning patients.

Conversely, the retrospective arm included all infertile couples initiating treatment between January 2012 and December 2021 at the Fertility Center. Data encompassing personal history and demographic details were extracted from the internal database of Humanitas Fertility Center to assess the factors involved in a treatment discontinuation.

Furthermore, all collected data were anonymized and all patients signed an informed consent to use their data for research purposes. A univariate analysis was performed to compare characteristics between returning and non-returning couples.

ELIGIBILITY:
Inclusion Criteria:

* The prospective study focused on patients discontinuing treatment following their initial visit to the Fertility Center of Humanitas Research Hospital, situated in Rozzano (Milan), Italy in 2021. These individuals were contacted by our staff and provided with a specific questionnaire via phone call.
* Conversely, the retrospective arm included all infertile couples initiating treatment between January 2012 and December 2021 at the same Center.

Exclusion Criteria:

* Excluded from our analysis were women not seeking conception.

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All infertile couples who had their first access at the Fertility Center of Humanitas Research Hospital, situated in Rozzano (Milan), Italy, between January 2012 and December 2021.
Sampling Method: Non-Probability Sample
Enrollment: 24773 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Dropout rate | 10 years
  The primary objective of this study was to determine the dropout rate of infertile couples after their first access to Humanitas Fertility Center.

SECONDARY OUTCOMES:
Reasons for dropout collected by a phone call questionnaire | 10 years
  Secondary aim was to assess the determinants in infertile couples influencing their choice not to return.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Emanuele Levi Setti, Study Director — Humanitas Research Hospital IRCCS, Rozzano-Milan
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No
Only under request

REFERENCES:
- [Derived] Scognamiglio C, Cirillo F, Ronchetti C, Secchi M, Busnelli A, Morenghi E, Alviggi C, Levi-Setti PE. From hope to hesitation: why couples fail to return for infertility treatment after the first consultation. Hum Reprod. 2025 May 1;40(5):919-925. doi: 10.1093/humrep/deaf012. PMID 40096631